CLINICAL TRIAL: NCT05944653
Title: Effects of the Interaction Between Physical Activity Level and Hormonal Status on Energy Metabolism and Nutritional Responses in Women
Brief Title: Physical Activity Level and Hormonal Status on Energy Metabolism and Nutritional Responses
Acronym: COCONUT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2023 DUCLOS; 2023-A00685-40 (Other: ANSM)
Record Dates: First submitted 2023-06-14; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Women; Metabolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with hormonal contraception
- Women without hormonal contraception

SUMMARY:
Obesity and its associated cardiometabolic comorbidities are a major health problem and although their prevalence is increasing in both men and women, evidence shows a faster increase in women, especially in those of childbearing age. In the scientific literature, cardiometabolic risks in women are often considered at menopause, younger women being considered "preserved" or less at risk than men. However, epidemiological studies show that it is essential to study and take into account these risks well before menopause, in particular in women of childbearing age, for their health but also for the health of future generations, considering the intergenerational cycle of women. However, the majority of studies have many limitations concerning the health of women of childbearing age since, in particular, they do not consider the hormonal and therefore physiological specificities of women. Indeed, the natural hormonal variations associated with the menstrual cycle but also the use of hormonal contraception, containing synthetic hormones, are important physiological modulators of these metabolic and nutritional regulations. Interestingly, in a recent narrative review, the investigators pointed out the little existing and reliable data concerning the effect of using oral contraception on the two sides of the energy balance, namely energy expenditure and energy intake. Also, it remains difficult to fully understand these metabolic and nutritional responses and therefore to optimize, whether in terms of primary or tertiary prevention, the health of women. Women using oral contraceptives activated the same brain pathways in response to food stimuli as women without contraception during the luteal phase, whereas these activations differed with respect to the follicular phase. Interestingly, women with overweight or obesity showed similar effects in terms of weight loss in response to an intervention including calorie restriction, a physical activity program and psychological support in women with and without hormonal contraception. However, while women without hormonal contraception managed to maintain the lost weight, women with contraception had a significant weight gain mainly due to an increase in their food intake. Conversely, in young healthy women following a calorie restriction of 500 kcal per week for one month, women with hormonal contraception showed greater weight loss than those without. Several parameters can potentially explain these differences in results, such as weight status, but also the nature of the intervention (i.e. caloric restriction only vs combined energy restriction and physical activity).

It is indeed recognized that the level of physical activity and sedentary behaviours influence the energy expenditure of rest and exercise and also the control of appetite; the investigators have recently shown that this level of physical activity modifies the cardiometabolic responses following a meal in healthy men. This underlines the importance of considering inter-individual parameters, such as the level of physical activity and sedentary lifestyle as a predominant factor in nutritional and energy regulation at rest and during physical exercise, a key factor in energy regulation. In general, studies in women concerning the parameters of the energy balance are heterogeneous in terms of the characteristics of the population, the methodology used and do not take into account all the metabolic and nutritional responses that make it possible to understand these regulations.

Thus, the main objective of this study is to evaluate the effects of hormonal status (women with and without hormonal contraception) on the fuel utilization during low-intensity physical exercise in women of childbearing age according to their level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 44y
* BMI between 18 and 25 kg.m-2
* Subject able to provide informed consent to participate
* Subject with a Social Security

Exclusion Criteria:

* Medical or surgical history judged by the investigator to be incompatible with the study
* Presence of comorbidities or pathology that could interfere with the study data
* Women in the process of food restriction or weight loss at the time of inclusion or during the last three months
* Irregular menstrual cycles
* Menstrual cycles < 25 days or greater than 35 days
* Pregnant or lactating women
* Per or post menopausal women
* Claustrophobia
* Person in period of exclusion from another study
* Person under guardianship or safeguard of justice; or subject without social security

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women with or without hormonal contraceptives
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory quotient | Through the 40 minute walking exercise
  It is the ratio of carbon dioxide production to oxygen consumption and represents the part of carbohydrate and fat oxidation

SECONDARY OUTCOMES:
Energy expenditure | Through the 40 minute walking exercise
  Oxygen consumption assessed by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France